CLINICAL TRIAL: NCT00257283
Title: A Double Blind Comparison of Omacor and Placebo as Secondary Prevention Against Cardiovascular Events in Patients Undergoing Chronic Hemodialysis
Brief Title: Omacor in Prevention of Cardiovascular Events in Patients Undergoing Chronic Hemodialysis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pronova BioPharma (Industry)
Collaborators: Danish Heart Foundation (Other); The Danish Kidney Association (Other); North Denmark Region (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CTN K85 02024
Record Dates: First submitted 2005-11-21; First posted 2005-11-22 (Estimated); Last update posted 2008-03-11 (Estimated); Status verified 2008-03

CONDITIONS: Kidney Failure, Chronic
Keywords: Chronic renal failure; Hemodialysis; OMACOR (omega-3-acid ethyl ester 90); intervention study; cardiovascular events; mortality
MeSH Terms: conditions — Kidney Failure, Chronic

INTERVENTIONS:
Drug: Omega-3-acid ethyl esters 90

SUMMARY:
The aim of this investigator initated study is to examine the effect of OMACOR (Omega-3-acid ethyl ester 90) on the incidence of cardiovascular events and mortality in patients undergoing chronic hemodialysis, who has previously experienced a cardiovascular event.

DETAILED DESCRIPTION:
Patients with renal failure have a high incidence of cardiovascular disease and increased premature mortality. Omega-3 polyunsaturated fatty acids from fish are known to have cardioprotective effects in subects with normal renal function. The aim of present study is to examine the effect of OMACOR (Omega-3-acid ethyl ester 90) on the incidence of cardiovascular events and mortality in patients undergoing chronic hemodialysis, who has previously experienced a cardiovascular event.

Design: A prospective, randomised, placebo controlled study. 2 year treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Males and females above 18 years of age
* Patients having been treated with chronic hemodialysis for at least 6 months
* Patients with documented cardiovascular disease, at least one of the following

  1. Angina pectoris
  2. Previous Acute myocardial infarction
  3. Previous PTCA/CABG or demonstated atheroclerosis after coronary angio
  4. Previous Transitory Cerebral Ischemia
  5. Previous Apoplexia Cerebri
  6. Symptoms of peripheral vascular disease
* Written informed consent

Exclusion Criteria:

* Active malignant disease, except basal cell carcinoma or spinocellular carcinoma
* Patients undergoing peritoneal dialysis
* Any condition associated with a risk of poor compliance, as judged by investigator
* Pregnant or breastfeeding
* Participation in other clinical studies involving treatment with drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2002-11; Study Completion 2005-06

PRIMARY OUTCOMES:
Composite endpoint, including either of the following events:
- Acute Myocardial Infarction
- Angina Pectoris, leading to coronary investigation or intervention
- Transient Cerebral Ischemia (TCI)
- Apoplexia cerebri (stroke)
- Peripheral Vascular disease, new symptoms or worsening of old symptoms
- Death

SECONDARY OUTCOMES:
- Efficacy laboratory variables (lipids, adhesion molecules, other efficacy lab variables, data for S-LDL-c size)
- Efficacy, fatty acid profile for phospholipids fraction
- Efficacy: diet registration, fish score
- Thrombosis and/or stenosis of dialysis graft
- Effect on heart rate variability, substudy of 50 patients at baseline and after three months

CONTACTS AND LOCATIONS:
Overall Officials: My Svensson, MD, Principal Investigator — Department of Nephrology, Aalborg Hospital, Aarhus University Hospital, Aalborg, Denmark
Locations (1):
- Department of Nephrology, Aalborg Hospital, Aarhus University Hospital, Aalborg, Denmark